CLINICAL TRIAL: NCT06938438
Title: Comparison of Single Locking Miniplates Versus Double Non-Locking Miniplates in Fixation of Anterior Mandibular Fracture
Brief Title: Single Locking Miniplates Versus Double Non-Locking Miniplates in Anterior Mandibular Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Maram Nashaat Breshah, Lecturer of Oral & Maxillofacial Surgery, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: #R-OS-2-22-12
Record Dates: First submitted 2025-04-14; First posted 2025-04-22 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2025-04

CONDITIONS: Anterior Mandibular Fracture
Keywords: anterior mandibular fracture; locking miniplate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: single locking miniplate (Active Comparator): Comprised of ten patients in whom anterior mandibular fractures will be fixed with titanium single locking miniplate
  Interventions: Procedure: single locking miniplate
- Group II: double conventional miniplates (Active Comparator): Comprised of ten patients in whom, anterior mandibular fractures will be fixed with double conventional titanium miniplates.
  Interventions: Procedure: double conventional miniplates.

INTERVENTIONS:
Procedure: single locking miniplate — Ten patients in whom anterior mandibular fractures will be fixed with titanium single locking miniplate
  Arms: Group I: single locking miniplate
Procedure: double conventional miniplates. — Ten patients in whom, anterior mandibular fractures will be fixed with double conventional titanium miniplates.
  Arms: Group II: double conventional miniplates

SUMMARY:
The aim of this study is to compare clinically and radiographically the using of single locking miniplate versus double non-locking miniplates in internal fixation of anterior mandibular fracture

DETAILED DESCRIPTION:
This study will be carried out on twenty adult patients with mandibular symphyeal and parasymphyseal fracture indicated for open reduction and internal fixation. The patients will be recieved, clinically& radiographically examined and managed at Oral & Maxillofacial Surgery Department, Faculty of Dentistry, Tanta University. Patients will be randomly divided into two equal groups according to the type of plating system used in fracture fixation: • Group I: Comprised of ten patients in whom anterior mandibular fractures will be fixed with titanium single locking miniplate. • Group II: Comprised of ten patients in whom, anterior mandibular fractures will be fixed with double conventional titanium miniplates.

Preoperative evaluation:

A thorough clinical examination will be performed for all patients.An intraoral clinical examination will be done to evaluate occlusal status, hematoma, soft tissue laceration, infection and neural disorder. Preoperative radiographic evaluation will be performed including standardized orthopantomograms (OPG) and CT radiographs to document the presence of the fracture and to determine the degree of displacement

Surgical Technique:

The patients will be operated under inhalational type of general anaesthesia via nasoendotracheal intubation. Disinfection of the surgical field with Betadine and surgical draping, Erich's arch bars will be applied. Mentalis muscle will be exposed and incised perpendicular and deep to the bone, leaving a flap of muscle attached to bone for closure. The mucoperiosteal flap will be raised.

In group I:

Adequate exposure of the fractured segments and adequate reduction of segments by manual reduction which assured by accurate occlusion and disappearance of step between segments. Once occlusion is achieved through intermaxillary fixation, five hole straight single locking titanium miniplate

In group II:

According to Champy principle two miniplates will be placed on the inferior border of the mandible and subapically will be used to fix fracture respectively.

Postoperative evaluation:

All patients of both groups will be evaluated clinically immediately, one week, two weeks, three weeks, four weeks, six weeks, three months and six months post-operatively regarding soft tissue healing, pain, edema, paraesthesia of lower lip, occlusion, stability of the fractured segments and Incidence of hardware failure.

Radiographic evaluation:

All patients will be evaluated using panoramic x-ray immediately and six months post-operatively. Axial, coronal and 3D CT scan will be done immediately and six months post-operatively. Immediate post-operative panoramic x-ray & CT scan will be done to display the fracture reduction and and the position of plate at the inferior border. Evaluation of bone healing at the fracture site and hardware failure and intergonial distance

ELIGIBILITY:
Inclusion Criteria:

* Patients with displaced symphyseal/ parasymphyseal mandibular fracture
* age group between 17-40 years old

Exclusion Criteria:

* Patients with systemic diseases that may affect bone healing
* Comminuted mandibular fracture.
* Edentulous patients

Ages: 17 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-09-20 (Actual)

PRIMARY OUTCOMES:
Soft tissue healing | 1 month
  either normal healing or dehiscence.
visual analogue scale | 1 month
  0 representing no pain at all and 10 representing severe pain
Edema | 1 month
  utilizing a horizontal and vertical guide with a tape on four reference points:tragus of the ear, soft tissue pogonion, pupil and the intersection between lines drawn from pupil centre falling vertically to inferior border of mandible and line parallel to inferior border of the mandible respectively then obtain the percentage of facial swelling, the difference between measurements of the postoperative and preoperative periods was divided by the value of the preoperative period.
Paraesthesia of lower lip | 6 months
  Two point discrimination test:
  Score 0: patients could not tell which tip was felt, even if these were morethan 20 mm apart.
  Score 1: patients could distinguish between tips only when the caliper wascalibrated at between 14 and 20 mm.
  Score 2: normal sensitivity, patients could discriminate between the tips at ashorter distance than 14 mm.
Occlusion | 6 months
  Uglesic's questionnaire 1. Evaluation of the occlusion after fracture treatment
  * 5 points: occlusion altered bilaterally.
  * 3 points: occlusion altered on one side .
    1 point: occlusion altered on one side. occlusal adjustment required. 3points: occlusion adequate on both sides but not the same as before injury. 5 points: good occlusion obtained 2. Self-evaluation of chewing after treatment
  * 5 points: not able to chew 0 points: on soft diet 3 points: on normal diet, but can chew only on one side 5 points: on normal diet
Stability of the fractured segments | 6 months
  stable/unstable based on clinical evaluation by digital palpation, applying pressure across fractured segments
bone healing at the fracture site | 6 months
  The fracture line could or could not be identified on radiograph
hardware failure | 6 months
  either plate fracture or screw loosening
Intergonial distance | 6 months
  Linear measurement by C.T software

CONTACTS AND LOCATIONS:
Overall Officials: Nesreen M Ramadan, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Mohamed M Shoushan, Prof, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Mohamed E Kamal, Ass Prof, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt; Maram N Breshah, Lecturer, Principal Investigator — Faculty of Dentistry, Tanta University, Egypt
Locations (1):
- Faculty of Dentistry, Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No